CLINICAL TRIAL: NCT01748084
Title: Evaluation of Rituximab in Systemic Sclerosis Associated Polyarthritis
Brief Title: Rituximab in Systemic Sclerosis
Acronym: RECOVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P110110; 2012-001636-56 (EudraCT Number)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Arthritis; B-cell therapy, Anti-CD20 therapy; Quality of life; Scleroderma; Lung fibrosis; Randomised controled trial
MeSH Terms: conditions — Scleroderma, Systemic; Arthritis; Scleroderma, Diffuse; Pulmonary Fibrosis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaCl (Placebo Comparator): NaCl 500 ml IV day 1 and day 15 plus 100 mg methylprednisolone
  Interventions: Drug: Placebo (NaCl)
- Rituximab (Experimental): Rituximab 1G IV day 1 and day 15 plus 100 mg methylprednisolone
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Days 1 and 15, rituximab 1 gramme plus 100 mg methylprednisolone
  Arms: Rituximab
Drug: Placebo (NaCl) — Days 1 and 15, NaCl 500 ml plus 100 mg methylprednisolone
  Arms: NaCl

SUMMARY:
The purpose of this study is to determine whether rituximab is effective in the treatment of articular symptoms that occur in systemic sclerosis related polyarthritis

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare disease, characterized by microvascular and immunological changes promoting extra-cellular matrix synthesis and widespread fibrosis. No treatment has yet proven any ability to alter the disease fibrosing process. Specific auto-antibodies are commonly found in this disease, and B lymphocytes are detected in cutaneous and pulmonary infiltrates. Studies derived from murine models suggest a role for B lymphocyte blocking strategies.

This lead to observational trials of B-cell therapy using rituximab in SSc that provided encouraging results with no particular signal concerning tolerability. These trials included heterogeneous patients with variable disease stages and different involved organs, and were mostly unblinded, which preclude any definitive conclusion. However, they support the continuous development of this therapeutic approach.

Taking up the early phase of the diffuse form of the disease is complicated by its rarity and the heterogeneous progression of its visceral complications. This raises the question of selecting a homogeneous group of patients to evaluate. The most convincing results for the use of rituximab in autoimmune conditions have been found in rheumatoid arthritis. Joint involvement is common in SSc with 75% of patients complaining about joint stiffness and pain, and 30% presenting with synovitis, tenosynovitis, or flexion contractures. No specific treatment has already addressed this issue, and it is generally proposed to use small doses of oral corticosteroids in association with methotrexate, by analogy with rheumatoid arthritis. We propose to evaluate the efficacy and safety of rituximab in SSc patients having active arthritis despite first line treatment. Improving the articular involvement would improve the quality of life f SSc patients and effectiveness of rituximab on skin and lung fibrotic involvements will be assessed as secondary outcomes to estimate the overall effects of this drug on SSc.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis fulfilling ACR or LeRoy's criteria
* Active polyarthritis defined by > 6/53 tender joints and > 4/53 swollen joints
* Ongoing first line therapy by prednisone (max 10 mg/d) and DMARDS (methotrexate, leflunomide, azathioprine or mycophenolate)
* Birth control if applicable

Exclusion Criteria:

* Overlap syndrome defined by clinical symptoms and positive specific auto-antibodies (anti-CCP, anti-SSA, anti-DNA DNA anti-Sm) (Rheumatoid factors and anti-RNP are not exclusion criteria)
* Past therapy with Rituximab.
* Severe and uncontrolled disease with renal, liver or haematological (neutropenia < 1500 / mm3) failures, pulmonary (FVC < 50%) or cardiac insufficiencies (LVEF < 50%)
* Not stable corticosteroid therapy or cyclophosphamide use in the last 6 months
* Infectious risk : viral infections by B or C hepatitis or HIV, hypogammaglobulinemia (< 6 G/L), opportunistic infection or infection requiring IV antibiotics in the last 3 months.
* Neoplastic solid tumor in the last 5 years
* Drug or alcool abuses
* Receiving patient or having received a biotherapy (anti-TNF, abatacept or tocilizumab) in the last 3 months (possible inclusion beyond 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2016-04-18 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
Number of tender and swollen joints | at 6 months
  Measured out of 53 joints

SECONDARY OUTCOMES:
Quality of life: SSc-HAQ | at 6 and 12 months
  Validated scores
Scleroderma | at 6 and 12 months
  modified Rodnan skin score
Lung fibrosis | at 6 and 12 months
  Pulmonary functional tests
Quality of life: SF-36 | at 6 and 12 months
  Validated scores
Quality of life: Duruöz index | at 6 and 12 months
  Validated scores

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Allanore, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris, Université Paris Descartes
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Bosello S, De Santis M, Lama G, Spano C, Angelucci C, Tolusso B, Sica G, Ferraccioli G. B cell depletion in diffuse progressive systemic sclerosis: safety, skin score modification and IL-6 modulation in an up to thirty-six months follow-up open-label trial. Arthritis Res Ther. 2010;12(2):R54. doi: 10.1186/ar2965. Epub 2010 Mar 25. PMID 20338043
- [Background] Simms RW, Lafyatis R. Rituximab: a potential therapeutic advance in scleroderma: what is the evidence? Rheumatology (Oxford). 2010 Feb;49(2):201-2. doi: 10.1093/rheumatology/kep421. Epub 2009 Dec 23. No abstract available. PMID 20032221
- [Background] Daoussis D, Liossis SN, Tsamandas AC, Kalogeropoulou C, Kazantzi A, Korfiatis P, Yiannopoulos G, Andonopoulos AP. Is there a role for B-cell depletion as therapy for scleroderma? A case report and review of the literature. Semin Arthritis Rheum. 2010 Oct;40(2):127-36. doi: 10.1016/j.semarthrit.2009.09.003. Epub 2009 Dec 11. PMID 20004954
- [Background] Daoussis D, Liossis SN, Tsamandas AC, Kalogeropoulou C, Kazantzi A, Sirinian C, Karampetsou M, Yiannopoulos G, Andonopoulos AP. Experience with rituximab in scleroderma: results from a 1-year, proof-of-principle study. Rheumatology (Oxford). 2010 Feb;49(2):271-80. doi: 10.1093/rheumatology/kep093. Epub 2009 May 15. PMID 19447770
- [Background] Lafyatis R, Kissin E, York M, Farina G, Viger K, Fritzler MJ, Merkel PA, Simms RW. B cell depletion with rituximab in patients with diffuse cutaneous systemic sclerosis. Arthritis Rheum. 2009 Feb;60(2):578-83. doi: 10.1002/art.24249. PMID 19180481